CLINICAL TRIAL: NCT03826212
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Soybean Germ Extract on Decrease of Body Fat
Brief Title: Efficacy and Safety of Soybean Germ Extract on Decrease of Body Fat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NOVA-BF-SBG
Record Dates: First submitted 2019-01-23; First posted 2019-02-01 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soybean Germ Extract (Experimental): Soybean Germ Extract 1,600 mg/day for 12 weeks.
  Interventions: Dietary Supplement: Soybean Germ Extract
- Placebo (Placebo Comparator): Placebo 1,600 mg/day for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soybean Germ Extract — Soybean Germ Extract 1,600 mg/day for 12 weeks.
  Arms: Soybean Germ Extract
Dietary Supplement: Placebo — Placebo 1,600 mg/day for 12 weeks.
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Soybean germ extract on decrease of body fat

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. 80 subjects were randomly divided into Soybean germ extract 1,600 mg or placebo group. The investigators measured Body Fat Mass, Percent Body Fat, Fat Free Mass, weight, and body mass index, etc.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 65 years
* BMI 25~29.9 kg/m^2
* After fully hearing and fully understanding this clinical trials, those who agree to voluntarily decide to participate and to comply with the notice

Exclusion Criteria:

* Those who lost more than 10% of their weight within 3 months before the screening
* Those who take a product(body fat improvement health functional foods, birth control pills, steroids, female hormone) that affects your weight within 4 weeks prior to the screening
* Those with clinically significant severe cardiovascular, endocrine, immune, respiratory, liver, biliary, renal and urinary tract, neuropsychiatry, musculoskeletal, inflammatory and hematologic and gastrointestinal disorders
* Diabetic patients taking oral hypoglycemic agents or insulin (based on screening subjects)
* A person with a history of clinically significant hypersensitivity to soybeans
* Those who have received antipsychotic medication within 2 months before screening
* Anyone with substance abuse or suspicion
* Those who participated in other clinical trials within 3 months before screening
* Systolic Blood Pressure(SBP) 180 mmHg, Diastolic Blood Pressure(DBP) 110 mmHg or more
* Menopausal woman
* Laboratory test by show the following results

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breast feeding
* Those who doesn't accept the implementation of appropriate contraception of a childbearing woman
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes of body fat mass | Baseline and 12 week
  Body fat mass was measured in study baseline and 12 week

SECONDARY OUTCOMES:
Changes of percent body fat | Baseline and 12 week
  Measurement is made using dual energy X-ray absorptiometry (DEXA / Hologic Discovery, USA). Left arm, right arm, left leg, right leg, trunk, total will be report percent body fat in %.
Changes of fat free mass | Baseline and 12 week
  Measurement is made using dual energy X-ray absorptiometry (DEXA / Hologic Discovery, USA). Left arm, right arm, left leg, right leg, trunk, total will be report fat free mass in g.
Changes of Anthropometric indicate: body weight | Screening, baseline and 12 week
  Anthropometric indices were measured in study screening, baseline and 12 week. Body weight in kg.
Changes of Anthropometric indicate: body mass index | Screening, baseline and 12 week
  Anthropometric indices were measured in study screening, baseline and 12 week. Weight/height^2 will be report body mass index in kg/m^2.
Changes of Anthropometric indices: waist circumference, hip circumference | Screening, baseline and 12 week
  Anthropometric indices were measured in study screening, baseline and 12 week. Waist circumference, hip circumference in cm.
Changes of Anthropometric indicate: waist -hip circumference ratio | Screening, baseline and 12 week
  Anthropometric indices were measured in study screening, baseline and 12 week. Waist circumference/hip circumference will be report waist -hip circumference ratio.
Changes of lipid metabolism indicators: Total cholesterol, Triglyceride, LDL-cholesterol, HDL-cholesterol | Baseline and 12 week
  Lipid metabolism indicators(mg/dL) were measured in study baseline and 12 week.
Changes of obesity-related hormones indicators: Adiponectin, Leptin | Baseline and 12 week
  obesity-related hormones indicators were measured in study baseline and 12 week
Changes of energy expenditure Indicators: Uncoupling protein-1(UCP-1), Peroxisome proliferator-activated receptor gamma coactivator-1 α(PGC-1 α) | Baseline and 12 week
  energy expenditure Indicators were measured in study baseline and 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea